CLINICAL TRIAL: NCT05039242
Title: Effects of Kinesiotaping for Hands Function in Patients With Rheumatoid Arthritis
Brief Title: Effects of Kinesiotaping for Hands Function in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01071 Summyyia Ayaz
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; Kinesio Tape; hand strength; Metacarpophalangeal Joint
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group A(Conventional Physical Therapy) (Active Comparator): Balanced resistive hand exercise with use of physio hand ball squeezes
  Interventions: Other: Conventional Physical Therapy)
- Experimental Interventional Group B (I-Band Application of Kinesiotaping) (Experimental): Participants will receive exercise interventions as group A along with that the Kinesiotape, by using I application technique from proximal to distal on dorsum of hand and forearm.
  Interventions: Other: Kinesiotaping with I shaped application
- Experimental Interventional Group C (fan shaped Application of Kinesiotaping) (Experimental): Participants will receive exercise interventions as group A along with that the Kinesiotape will be applied, by using fan cut application technique on MCP joints involving extensor tendons of fingers on dorsal surface of both hands of subjects
  Interventions: Other: Kinesiotaping with Fan-shaped Application

INTERVENTIONS:
Other: Conventional Physical Therapy) — Participants will receive a Hand exercise program including 8 different movements according to Flat 20 (flexion, extension, radial deviation of the fingers, dorsal flexion, palmar flexion, ulnar deviation of the fingers, and opposition and abduction of thumbs.
  Repetitions include 5 times during each session, as given in the study. Balanced resistive hand exercise with use of physio hand ball squeezes including finger abduction and adduction exercises with MCP extended and gross grip.
  Each contraction to be held for 3-5 seconds with a 20-second rest between contractions. Five repetitions of each resistive exercise will be done.
  Arms: Control Group A(Conventional Physical Therapy)
Other: Kinesiotaping with I shaped application — Participants will receive Kinesiotape, by using I application technique from proximal to distal on dorsum of hand and forearm with less than 50% stretch of the subjects on both hands, once a week for a total time period of 4 weeks with 4 KT applications in total (19). Kinesiotape will be worn by the subjects for 3 days. basic hand exercises will accompny it. Weekly assessments will be completed for pain, ROM, joint stiffness, grip strength and ADLs.
  Arms: Experimental Interventional Group B (I-Band Application of Kinesiotaping)
Other: Kinesiotaping with Fan-shaped Application — Participants will receive exercise interventions as group A along with that the Kinesiotape will be applied, by using fan cut application technique on MCP joints involving extensor tendons of fingers on dorsal surface of both hands of subjects, once a week for a total time period of 4 weeks with 4 KT applications in total.
  Kinesiotape will be worn by the subjects for 3 days. Less than 50% stretch with space correction technique. basic hand exercises will accompny it. Weekly assessments will be completed for pain, ROM, joint stiffness, grip strength and ADLs.
  Arms: Experimental Interventional Group C (fan shaped Application of Kinesiotaping)

SUMMARY:
The aim of this research is to compare the effects of I-shape and fan shape kinesiotape techniques on pain, range of motion, grip strength and ADLs of patients with Rheumatoid Arthritis. Randomized controlled trials done at Pain Clinic, Rawalpindi and Fauji Foundation Hospital, Rawalpindi. The sample size was 66. The subjects were divided in three groups, 22 subjects in control group receiving conventional physical therapy treatment, 22 subjects in second group with I-Band application of kinesiotaping and 22 in the third group with fan-shaped application of kinesiotaping. Study duration was of 6 months. Sampling technique applied was non-probability convenience sampling. Only 25-50 years symptomatic female patients with established RA were included. Tools used in the study are Michigan Hand Outcome Questionnaire (MHQ), Numeric Pain Raiting Scale, Dynamometer and Goniometer. Data was be analyzed through SPSS 21.

DETAILED DESCRIPTION:
Rheumatoid Arthritis is an autoimmune systemic condition characterized by joint inflammation and extra-articular erosions. The symptoms of RA usually progress with age from mild to severe. The progression can either occur insidiously over a period of months or it can occur in weeks or overnight. RA with symptoms lasting less than six months is called as "early", while with symptoms lasting longer than this is known as "established". RA has significant direct costs, such as health-care costs, as well as indirect costs, such as lost income due to morbidity and reduced life expectancy. In the urban population of southern Pakistan, Karachi, the prevalence of RA is reported to be 0.142%, whereas in northern Pakistan the estimated prevalence is 0.55%. In 2014, the overall age-adjusted prevalence of RA ranged from 0.53 to 0.55% (0.29-0.31% for males and 0.73-0.78% for females). In general, rheumatoid arthritis preferentially affects women with female to male ratio of about 3:1; however, patients with above 60 years of age have equal female to male ratio. The most prevalent age is 45-60 years. The disease severity increases with increase in the age and reaches to its peak in above 60 years of age.

The joints of hand affected by of RA include polyarthritis of small joints like proximal interphalengeal (PIP), metacarpophalengeal (MCP) joints, wrist and metatarsophalangeal (MTP) joints. Patients experience morning stiffness in these joints which lasts unto several hours. The signs on examination involves swelling, stiffness, tenderness over the affected joints, decreased range of motion and deformity like; trigger finger, boutonniere and swan neck deformity. These signs results in loss of function and mobility. Moreover, the progression of RA occurs in four stages. Stage 1 has no destructive changes on x-ray, stage 2 shows periarticular osteoporosis and subchondral bone destruction on x-ray with no joint deformity, stage 3 reveals periarticular osteoporosis with cartilage and bone destruction on x-ray and significant joint deformity and stage 4 proceeds with stage 3 with the addition of bony and fibrous ankylosis Rheumatoid arthritis is a chronic, incurable disease. All of the currently known treatments are aimed at alleviating symptoms and increasing quality of life. Treatments aim to relieve pain and decrease the progression of RA in order to prevent disability and improve functional capability . The four most common components of Physical therapy for RA hands are exercise therapy, joint protection advice and provision of functional splinting and assistive devices, massage therapy and patient education. Exercise therapy includes ROM exercises, aerobic exercise and stabilization/coordination exercises. Joint protection includes rest and splinting that uses orthosis to prevent the development of deformities and support joints. Massage therapy involves manual trigger of an articular movement focused on the improvement of function, pain reduction, reduction of disease activity improve flexibility and welfare (dimension of depression, anxiety, mood and pain). Patient education is done to inform them about their disease and the various therapies available to help them live a better life. Additional interventional strategies include application of cold therapy, heat therapy, Transcutaneous Electrical Nerve Stimulation (TENS) and hydrotherapy exercises are also beneficial as they induce minimal loads on the joints during exercise.

In 2016 Sarah Roberts et al conducted an RCT in order to check the effects of kinesio tape on pain and metacarpophalengeal joints of hands in patients with rheumatoid arthritis, the results revealed significant reduction in pain, improvement in ROM and enhanced grip strength in work and ADLs. Another study in 2016 conducted by Vilija Zebrauskaite et al in their study about the additive effects of kinesiotape for physiotherapy of patients with rheumatoid hand to correct to ulnar positioning of hand and improve hand function. The results were significantly positive with the hand function improved considerably in comparison with the group receiving only physiotherapy exercises. In 2019 Majid Farhadian et al conducted an RCT to investigate the effects of kinesio tape on pain, range of motion, hand strength and functional abilities in patients with hand osteoarthritis. The findings of this study revealed that Kinesio taping and hand training may help patients with HOA improve their discomfort, range of motion, hand strength, and upper-extremity functional capacities. Furthermore, these two approaches can be utilised in conjunction for the treatment of this illness.

The previous studies have shown the positive effects of kinesiotape on hand functions of patients with RA. Since kinesiotape has vast variety of application techniques, and in order to determine the effectiveness of each application technique, current study is going to be conducted to compare the effects of I strip application technique and fan cut or web strip application technique.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic subjects having age between 18-60 years.
* Patients with diagnosed established Rheumatoid Arthritis of Hands (i.e greater than 6 months of onset of Rheumatoid Arthritis).
* Patients who are currently experiencing pain in their hands.

Exclusion Criteria:

* Patients with any malignancy, infections, open wounds, skin allergy, cellulitis, DVT or any deformities of hands.
* Patients with co-morbidities including congestive heart failure, kidney disease, or any neurological deficits.
* Patients with other conditions affecting hands except Rheumatoid Arthritis.
* Patients with any history of hand surgery.
* Patients not presenting for follow up on designated date (every 6th day)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Score | 4th week
  The NPRS is used to measure the the pain at metacarpoplaalngeal joints. its a11- point scale with 0 showing no pain and 10 showing maximum pain
hand strength | 4th week
  hand strength is measured by dynamometer. the person grips the dynamometer and the reading shows the hand and grip strength

SECONDARY OUTCOMES:
metacarpoplahangeal Flexion Rt hand | 4th week
  the flexion ROM will be measured by the goniometer.
metacarpoplahangeal Extension Rt hand | 4th week
  the extension ROM will be measured by the goniometer.
metacarpoplahangeal flexion Lt hand | 4th week
  the flexion ROM will be measured by the goniometer.
metacarpoplahangeal Extension Lt hand | 4th week
  theExtension ROM will be measured by the goniometer.
wrist Extension Rt hand | 4th week
  the Extension ROM will be measured by the goniometer.
wrist Flexion Rt hand | 4th week
  the Flexion ROM will be measured by the goniometer.
ulnar deviation Rt hand | 4th week
  the ulnar deviation ROM will be measured by the goniometer.
radial deviation Rt hand | 4th week
  the radial deviation ROM will be measured by the goniometer.
wrist Extension Lt hand | 4th week
  the Extension ROM will be measured by the goniometer.
wrist Flexion Lt hand | 4th week
  the Flexion ROM will be measured by the goniometer.
ulnar deviation Lt hand | 4th week
  the ulnar deviation ROM will be measured by the goniometer.
radial deviation Lt hand | 4th week
  the radial deviation ROM will be measured by the goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- fouji Foundation hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chauhan K, Jandu JS, Goyal A, Bansal P, Al-Dhahir MA. Acute Rheumatoid Arthritis.
- [Background] Ottawa Panel. Ottawa Panel evidence-based clinical practice guidelines for therapeutic exercises in the management of rheumatoid arthritis in adults. Phys Ther. 2004 Oct;84(10):934-72. PMID 15449978
- [Background] Alam SM, Kidwai AA, Jafri SR, Qureshi BM, Sami A, Qureshi HH, Mirza H. Epidemiology of rheumatoid arthritis in a tertiary care unit, Karachi, Pakistan. J Pak Med Assoc. 2011 Feb;61(2):123-6. PMID 21375157
- [Background] Hunter TM, Boytsov NN, Zhang X, Schroeder K, Michaud K, Araujo AB. Prevalence of rheumatoid arthritis in the United States adult population in healthcare claims databases, 2004-2014. Rheumatol Int. 2017 Sep;37(9):1551-1557. doi: 10.1007/s00296-017-3726-1. Epub 2017 Apr 28. PMID 28455559
- [Background] Jalil F, Arshad M, Bhatti A, Jamal M, Ahmed M, Malik JM, Ali S, Akbar F, John P. Progression pattern of rheumatoid arthritis: A study of 500 Pakistani patients. Pak J Pharm Sci. 2017 Jul;30(4):1219-1223. PMID 29039317
- [Background] Williams MA, Williamson EM, Heine PJ, Nichols V, Glover MJ, Dritsaki M, Adams J, Dosanjh S, Underwood M, Rahman A, McConkey C, Lord J, Lamb SE. Strengthening And stretching for Rheumatoid Arthritis of the Hand (SARAH). A randomised controlled trial and economic evaluation. Health Technol Assess. 2015 Mar;19(19):1-222. doi: 10.3310/hta19190. PMID 25748549
- [Background] Dakkak YJ, Jansen FP, DeRuiter MC, Reijnierse M, van der Helm-van Mil AHM. Rheumatoid Arthritis and Tenosynovitis at the Metatarsophalangeal Joints: An Anatomic and MRI Study of the Forefoot Tendon Sheaths. Radiology. 2020 Apr;295(1):146-154. doi: 10.1148/radiol.2020191725. Epub 2020 Feb 11. PMID 32043949
- [Background] Walters JE, Brown AR, Jones AE. Use of the Copenhagen Burnout Inventory with social workers: a confirmatory factor analysis. Human Service Organizations: Management, Leadership & Governance. 2018;42(5):437-56.
- [Background] Williams MA, Srikesavan C, Heine PJ, Bruce J, Brosseau L, Hoxey-Thomas N, Lamb SE. Exercise for rheumatoid arthritis of the hand. Cochrane Database Syst Rev. 2018 Jul 31;7(7):CD003832. doi: 10.1002/14651858.CD003832.pub3. PMID 30063798
- [Background] de Jong Z, Munneke M, Zwinderman AH, Kroon HM, Jansen A, Ronday KH, van Schaardenburg D, Dijkmans BA, Van den Ende CH, Breedveld FC, Vliet Vlieland TP, Hazes JM. Is a long-term high-intensity exercise program effective and safe in patients with rheumatoid arthritis? Results of a randomized controlled trial. Arthritis Rheum. 2003 Sep;48(9):2415-24. doi: 10.1002/art.11216. PMID 13130460